CLINICAL TRIAL: NCT06007053
Title: Retraining and Control Therapy (ReACT): Sense of Control and Catastrophic Symptom Expectations as Targets of a Cognitive Behavioral Treatment for Pediatric Psychogenic Non-epileptic Seizures (PNES) - R33 Phase
Brief Title: Retraining and Control Therapy (ReACT) R33 Phase
Acronym: ReACT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Aaron Fobian, Associate Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB-151001004
Record Dates: First submitted 2023-08-11; First posted 2023-08-23 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Convulsion, Non-Epileptic
Keywords: Supportive therapy; ReACT
MeSH Terms: conditions — Seizures | interventions — Palliative Care

STUDY DESIGN:
Intervention Model Description: Children with PNES and matched controls will be prospectively enrolled. PNES participants will be randomized to either supportive therapy or Retraining and Control Therapy (ReACT).
Who Masked: Investigator, Outcomes Assessor
Masking Description: Researchers who conduct baseline and follow-up visits will be blinded to the condition to which the patient has been assigned. The statistician and data manger will be blinded to treatment condition when analyzing data. The PI and therapists will be blinded to participant's baseline target scores.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ReACT Intervention (Experimental): At the end of the baseline visit, half of the participants will be randomized to receive Retraining and Control Therapy (ReACT)
  Interventions: Behavioral: ReACT
- Supportive Therapy (Active Comparator): At the end of the baseline visit, half of the participants will be randomized to receive supportive therapy
  Interventions: Behavioral: Supportive Therapy
- Healthy Control (No Intervention): Healthy controls are ages 12-18 with no significant comorbid medical or mental health conditions. Healthy controls and their parent come for 1 baseline laboratory visit and a follow up visit 13 weeks after the baseline visit. These visits will be identical to baseline and follow-up visits of children with PNES.

INTERVENTIONS:
Behavioral: ReACT — ReACT is a novel cognitive behavioral treatment and is a PNES intervention that targets sense of control and catastrophic symptom expectations. ReACT consists of 12 sessions of therapy focused on teaching adolescents to regain control of their body through managing thoughts and behaviors that reinforce the PNES and return to previous activities. It teaches parents how to respond to PNES in a manner that encourages the adolescents to regain control of their body. The PNES is explained as behaviors learned through classical and operant conditioning.
  Other Names: Retraining and Control Therapy
  Arms: ReACT Intervention
Behavioral: Supportive Therapy — The supportive therapy treatment consists of 12 sessions of therapy focused on discussing daily difficulties and/or stressors they experience and identifying stress triggers for PNES. The PNES is explained as physical manifestations of psychological stress.
  Arms: Supportive Therapy

SUMMARY:
The purpose of this study is to assess sense of control and catastrophic symptom expectations as targets for Retraining and Control Therapy (ReACT- an intervention focused on changing behaviors and thoughts) for treatment of pediatric psychogenic non-epileptic seizures (PNES, episodes resembling epileptic seizures but with no correlated epileptiform activity). 11-18-year-olds diagnosed with PNES will engage in twelve sessions of either ReACT or supportive therapy. Sense of control over actions will be measured by the magic and turbulence task, a well-validated measure of sense of control. Participants will complete the cold pressor test (CPT) in which participants hold their hand in cool water for as long as possible up to 3 minutes. Catastrophic symptom expectations in response to the CPT will be measured by Pain Catastrophizing Scale for Children (PCS-C), pain tolerance (time with hand in water) and cortisol response. Target assessments occur 7 days before treatment, 7 days after 12th treatment session, and 2 months after the 12th treatment session. Long term follow-up assessments will occur 6 months and 12 months after the 12th treatment session. PNES frequency will be measured from 30 days before to 12 months after treatment.

DETAILED DESCRIPTION:
Participants with PNES and their parent come to our laboratory for a baseline visit and 4 follow-up visits. After the baseline visit, participants are randomized to 12 sessions of either Retraining and Control Therapy (ReACT) or supportive therapy. The first therapy session is in-person, and the following 11 sessions are completed via telehealth.

During the baseline visit, participants and their parent complete several questionnaires assessing demographics, mood and suicidality, relationships with friends and family, as well as past and current PNES symptoms. They also complete the childhood trauma questionnaire. The treatment targets (sense of control and catastrophic symptom expectations) are measured by the magic and turbulence computer task and pain tolerance, PCS-C and cortisol response to the CPT, respectively. PNES diaries are completed to assess PNES frequency over the previous 30 days. The baseline lab visit lasts about 2.5 hours. Saliva is collected over 1 time point before and 3 time points after the CPT to measure cortisol response to the CPT. Participants also collect 2 saliva samples 24 hours later to serve as a baseline outside of the laboratory setting. Participants will also be given a Respironics Actiwatch Spectrum Pro to track sleep and PNES episode severity and frequency for the 1 week between the baseline visit and first therapy session.

After the baseline visit, participants are scheduled to return in one week for their first of 12 intervention sessions of either ReACT or supportive therapy. This first session lasts a maximum of two hours, and the following 11 sessions are scheduled weekly and last one hour. The following 11 sessions are conducted as telehealth visits via HIPAA-compliant Zoom. Before beginning the first ReACT session, participants will complete the Flanker Inhibitory Control and Attention, List Sorting Working Memory, Pattern Comparison Processing Speed, Dimensional Change Card Sort, and Picture Sequence Memory subtests. Participants will be mailed another Respironics Actiwatch Spectrum Pro before the 11th therapy session to track sleep and PNES episode severity and frequency for the 2 weeks between the 11th therapy session and the lab visit one week after the 12th treatment session.

Follow-up at 7 days after treatment and 2 months after treatment also is conducted to perform tasks and complete follow-up assessment of the targets (sense of control and catastrophic symptom expectations), PNES frequency, and questionnaires. Each of these sessions last 2 hours. Participants will complete the Flanker Inhibitory Control and Attention, List Sorting Working Memory, Pattern Comparison Processing Speed, Dimensional Change Card Sort, and Picture Sequence Memory subtests at the lab visit at each of these visits. Participants will be mailed and asked to collect 2 saliva samples 1 day before they come in for their follow-up lab visit occuring 7 days after treatment. Participcants will complete 2 Zoom visits at 6 months and 12 months after treatment to assess long-term PNES outcomes and questionnaire data. These appointments will last 1 hour. PNES frequency will be measured from 30 days before treatment to 12 months after treatment through PNES diaries completed by the parent and the participant.

Participants will be offered the treatment to which they were not randomized after the 2-month follow-up when the study is completed.

After treatment, booster therapy sessions will be offered as needed.

Healthy controls will be recruited. Healthy controls and their parent come for a baseline laboratory visit and a follow up visit 13 weeks after the baseline visit. The baseline and follow-up appointments for healthy controls will be identical to the visits for children with PNES.

ELIGIBILITY:
Inclusion Criteria:

* 11-18 years old.
* Diagnosis of psychogenic non-epileptic seizures by a medical doctor using video-EEG.
* Family member (parent/guardian if a minor) willing to participate and that the subject with PNES chooses.

Exclusion Criteria:

* Comorbid Epilepsy
* Less than 4 PNES per month
* Other paroxysmal nonepileptic events (e.g. episodes related to hypoxic-ischemic phenomena, sleep disorders or migraine-associated disorders)
* Participation in other therapy during the study
* Severe intellectual disability
* Severe mental illness (delusions/hallucinations)

Exclusion for CPT:

* Blood pressure >130/80 mmHg for adolescents greater than or equal to 13 years old
* Either systolic and/or diastolic blood pressure greater than or equal to 95% based on sex and age for children less than 13 years old

Ages: 11 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 160 (Estimated)
Dates: Start 2024-03-09 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Magic and turbulence task | 7 months
  Measure of perceived sense of control in response to tasks in which control is manipulated; Greater negative numbers indicate improved understanding of control. Assessed at baseline visit, and 1 week and 2 months after the final therapy sessions (about 7 months total).
Pain catastrophizing scale for children- situation specific | 7 months
  Measures catastrophic symptom expectations; score ranges from 0-52, higher scores indicate greater levels of pain-related anxiety. Assessment done after performing Cold Pressor Test. Assessed at baseline visit, and 1 week and 2 months after the final therapy sessions (about 7 months total).
Pain tolerance (time) | 7 months
  Measures catastrophic symptom expectations. Measured by the total time the participant can keep their hand in cool water during the Cold Pressor Test. Shorter time indicates less pain tolerance. Assessed at baseline visit, and 1 week and 2 months after the final therapy sessions (about 7 months total).
Salivary Cortisol | 7 months
  Measures catastrophic symptom expectations. Measured before and after the cold pressor test. Increased cortisol response indicate increased perceived pain severity. Assessed at baseline visit, and 1 week and 2 months after the final therapy sessions (about 7 months total).
Pain Rating Scale | 7 months
  Measures perceived pain severity after the CPT; score ranges from 0-100. Higher scores indicate greater perceived pain severity. Assessed at baseline visit, and 1 week and 2 months after the final therapy sessions (about 7 months total).
Stroop task | 7 months
  Measure of cognitive inhibition and selective attention, higher scores means poorer cognitive inhibition and selective attention. Assessed at baseline visit, and 1 week and 2 months after the final therapy sessions (about 7 months total).

SECONDARY OUTCOMES:
PNES Frequency | 16 months
  Measured by Psychogenic Non-epileptic Seizures (PNES) diary, including frequency, premonitory symptoms, description of PNES symptoms and duration. Assessed 30 days before treatment to 12 months after the 12th treatment session (about 16 months total).
Pain Catastrophizing Scale for Children (PCS-C)- General | 7 months
  Measures catastrophic symptom expectations; score ranges from 0-52, higher scores indicate greater levels of pain-related anxiety. Assessment done before performing Cold Pressor Test. Assessed at baseline visit, and 1 week and 2 months after the final therapy sessions (about 7 months total).
Children's Somatic Symptoms Inventory (CSSI-24) | 16 months
  General somatic symptom complaints, higher scores indicate greater somatic complaints. Scores range from 0-140. Completed by participant and parent. Assessed at baseline visit, and 1 week, 2 months, 6 months and 12 months after the final therapy sessions (about 16 months total).
Anxiety Sensitivity Index (ASI) | 16 months
  Assesses catastrophic symptom expectations; scores ranges from 0-64, higher scores indicate greater anxiety. Completed by participant and parent. Assessed at baseline visit, and 1 week, 2 months, 6 months and 12 months after the final therapy sessions (about 16 months total).
Shipley | At Baseline
  Assesses verbal IQ; higher scores indicate greater verbal IQ. Completed by participant. Assessed at baseline visit.
Quality of Life in Epilepsy for Adolescents (QOLIE-AD-48) | 16 months
  Assesses health-related quality of life for children with epilepsy (used in PNES participants by instructing them to consider their PNES when asked about "seizures"); score ranges from 0-100, higher scores indicate better functioning and well-being. Completed by participant. Assessed at baseline visit, and 1 week, 2 months, 6 months and 12 months after the final therapy sessions (about 16 months total).
Sense of Agency Question | 16 months
  Single question which asks "How much control do you believe you have over your PNES?", scored using a 4-point Likert scale. Lower score indicates better control over PNES. Completed by participant. Assessed at baseline visit, and 1 week, 2 months, 6 months and 12 months after the final therapy sessions (about 16 months total).
LEVEL 2-Somatic Symptom report adapted from the Participant Health Questionnaire | 16 months
  Measures symptom severity in children; scores ranges from 0-26, higher scores indicate greater symptom severity. Completed by participant and parent. Assessed at baseline visit, and 1 week, 2 months, 6 months and 12 months after the final therapy sessions (about 16 months total).
Functional Disability Inventory (FDI) | 16 months
  Completed by child and parent to measure physical functioning and disability in children with chronic pain; score ranges from 0-60, higher scores indicate greater perceived functional disability. Completed by participant and parent. Assessed at baseline visit, and 1 week, 2 months, 6 months and 12 months after the final therapy sessions (about 16 months total).
The Impact on Family Scale | 16 months
  Assesses parental perceptions of the impact of a child's medical condition on the family; higher scores indicate greater financial burden on the family. Assessed at baseline visit, and 1 week, 2 months, 6 months and 12 months after the final therapy sessions (about 16 months total).
Childhood Trauma Questionnaire | At baseline
  History of physical, sexual and/or emotional abuse and physical and emotional neglect. All clinical subscales have a score range of 5-25, higher scores indicate greater abuse/neglect. Completed by participant. Assessed at baseline visit.
The Revised Children's Anxiety and Depression Scale (RCADS) | 16 months
  Measures anxiety and depression symptoms in children; total score ranges from 0-141, higher scores indicate increased symptom severity. Completed by participant and parent. Assessed at baseline visit, and 1 week, 2 months, 6 months and 12 months after the final therapy sessions (about 16 months total).
The Columbia Suicide Severity Rating Scale (C-SSRS) | 16 months
  Measure that addresses the full range of suicidal thoughts and behaviors that suggest a person is at heightened risk of committing suicide; score ranges from 0-25, higher score indicates greater suicidal ideation intensity. Completed by trained research study coordinator.Assessed at baseline visit, and 1 week, 2 months, 6 months and 12 months after the final therapy sessions (about 16 months total).
Healthcare Related Stigma Questionnaire | At Baseline
  Measures stigma in patients and their parents related to their interaction with health care; scores ranges from 0-64, higher scores indicate greater stigma. Completed by participant and parent. Assessed at baseline visit.
COVID-19 Functional Neurological Disorders (FND) Questionnaire | At Baseline
  Assesses the effect of COVID-19 diagnosis in FND patients (not on a rating scale). Completed by children. Assessed at baseline visit.
Flanker Inhibitory Control and Attention Subtest | 7 months
  Subtest of the National Institute of Health Toolbox Cognition Battery. Measures executive function and attention; higher scores indicate better performance. Completed by children. Assessed at 1st therapy session, and 1 week and 2 months after 12th therapy session (about 7 months total).
List Sorting Working Memory Subtest | 7 months
  Subtest of the National Institute of Health Toolbox Cognition Battery. Measures working memory; higher scores indicate better performance. Completed by children. Assessed at 1st therapy session, and 1 week and 2 months after 12th therapy session (about 7 months total).
Pattern Comparison Processing Speed Subtest | 7 months
  Subtest of the National Institute of Health Toolbox Cognition Battery. Measures processing speed; higher scores indicate better performance. Completed by children. Assessed at 1st therapy session, and 1 week and 2 months after 12th therapy session (about 7 months total).
Dimensional Change Card Sort Subtest | 7 months
  Subtest of the National Institute of Health Toolbox Cognition Battery. Measures executive function; higher scores indicate better performance. Completed by children. Assessed at 1st therapy session, and 1 week and 2 months after 12th therapy session (about 7 months total).
Picture Sequence Memory Subtest | 7 months
  Subtest of the National Institute of Health Toolbox Cognition Battery. Measures episodic memory; higher scores indicate better performance. Completed by children. Assessed at 1st therapy session, and 1 week and 2 months after 12th therapy session (about 7 months total).
Sleep Duration | 4 months
  Measures total sleep duration in a 24-hour day. Objectively measured using Respironics Actiwatch Spectrum Pro and subjectively measured using sleep diaries. Worn/completed by children. Assessed for 1 week between baseline visit and 1st therapy session and 2 weeks between 11th therapy session and 1 week after 12th therapy session (about 4 months total).
Sleep Efficiency | 4 months
  Measures quality of sleep. Objectively measured using Respironics Actiwatch Spectrum Pro and subjectively measured using sleep diaries. Worn/completed by children. Assessed for 1 week between baseline visit and 1st therapy session and 2 weeks between 11th therapy session and 1 week after 12th therapy session (about 4 months total).
Sleep Onset Latency | 4 months
  Refers to the time it took the child to fall asleep after lying down in bed. Objectively measured using Respironics Actiwatch Spectrum Pro and subjectively measured using sleep diaries. Worn/completed by children. Assessed for 1 week between baseline visit and 1st therapy session and 2 weeks between 11th therapy session and 1 week after 12th therapy session (about 4 months total).
Sleep - Bed Time | 5 months
  Measures total time in bed in a 24-hour day. Objectively measured using Respironics Actiwatch Spectrum Pro and subjectively measured using sleep diaries. Worn/completed by children. Assessed for 1 week between baseline visit and 1st therapy session and 2 weeks between 11th therapy session and 1 week after 12th therapy session (about 5 months total).
Sleep - Wake Time | 4 months
  Measures total awake time in a 24-hour day. Objectively measured using Respironics Actiwatch Spectrum Pro and subjectively measured using sleep diaries. Worn/completed by children. Assessed for 1 week between baseline visit and 1st therapy session and 2 weeks between 11th therapy session and 1 week after 12th therapy session (about 4 months total).
PNES Episode Frequency | 4 months
  Measures the total number of PNES episodes the child had in a day. Objectively measured using Respironics Actiwatch Spectrum Pro. Worn by children. Assessed for 1 week between baseline visit and 1st therapy session and 2 weeks between 11th therapy session and 1 week after 12th therapy session (about 4 months total).
PNES Episode Duration | 4 months
  Measures the duration of a PNES episode. Objectively measured using Respironics Actiwatch Spectrum Pro. Worn by children. Assessed for 1 week between baseline visit and 1st therapy session and 2 weeks between 11th therapy session and 1 week after 12th therapy session (about 4 months total).
Rosenberg Self-esteem scale | 16 months
  This is a 10-item scale measuring self esteem. Score ranges from 0-30 with low scores indicating low self-esteem. Completed by participant at baseline visit and follow-up visits.
Beaver's Self-Report Family Inventory | 16 months
  This is a 36 item scale which assesses a family member's view of overall family competence. Completed by participant at baseline visit. Completed by parent at baseline and follow-up visits.
FND Locus of Control: Multidimensional Health Locus of Control (MHLC) Scales | 16 months
  Measures an individual's belief in his/her ability to control health outcomes. Form C of MHLC scale will be completed by participant and Form A of MHLC scale will be completed by parent. Assessed at baseline visit and follow-up visits.
Dysfunctional Attitude Scale (DAS-9) | 16 months
  Participant will complete this 9-item self-report measure that aims to determine stable negative attitudes that people with depression hold about themselves, the world, and their future. Assessed at baseline visit and follow-up visits.
Mishel Uncertainty in Illness Questionnaire-Community Form (MUIS-C) | 16 months
  Participant will complete this 23-item scale which measures uncertainty about their diagnosis. Assessed at baseline visit and follow-up visits.
Parenting Style and Dimensions Questionnaire (PSDQ Short Version) | 5 to 7 months
  This is a 32-item scale assessing parenting style (self and spouse). Completed by parent at baseline visit and 7-day follow-up visit.
Revised Helping Alliance Questionnaire- II | 16 months
  Revised Helping Alliance Questionnaire-II is a 19-item scale will assess the therapist, children and parents' perception of the therapeutic alliance at follow-ups. Scores ranges from 19-114 with a higher score indicating better therapeutic alliance. Completed at baseline and follow-up visits.
The Credibility/Expectancy Questionnaire | 16 months
  The Credibility/Expectancy Questionnaire will be used to compare treatment expectancy between conditions. It measures how much the patient believes the therapy they are receiving will help to reduce their FS. This will be completed initially after being randomized, after the first session, fourth session, eighth session, and at the follow-up visits.
Session Summary Sheet (SSS) | 5 to 7 months
  Assesses parent and participant's therapeutic relationship, mastery of skill and involvement in therapy session. Completed by therapist at each intervention visit.
Illness Cognitions Scale | 16 months
  Participant will complete this 17-item scale measuring the degree to which they align with the sick role. Assessed at baseline visit and follow-up visits.
Other FND Symptoms Questionnaire | 16 months
  Assesses if participant has other functional symptoms (independent from their PNES), and evaluates the intensity and frequency of these symptoms. Completed by parent at Baseline and follow-up visits
Clinical Global Impression | 5 to 7 months
  Assesses the participant's improvement in FS/FND symptoms due to treatment intervention. Completed by therapist at every treatment session.

CONTACTS AND LOCATIONS:
Overall Officials: Aaron Fobian, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States